CLINICAL TRIAL: NCT02019446
Title: Evaluating the Effectiveness of Laser Treatment for Onychomycosis of the Hallux in Patients With Diabetes: A Randomized Controlled Trial
Brief Title: Laser Treatment for Onychomycosis in Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BCDiabetes.Ca (Network)
Collaborators: BritaMed, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H13-03369
Record Dates: First submitted 2013-12-16; First posted 2013-12-24 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2; Onychomycosis
Keywords: type 2 diabetes mellitus; onychomycosis; laser treatment; antifungal
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Onychomycosis | interventions — Control Groups; Terbinafine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Laser Treatment (Experimental): Participants randomized to laser group will undergo laser treatment at baseline and be asked to return for 2 subsequent visits six weeks apart (at weeks 6 and 12) to undergo further laser treatment of the hallux. Each visit will last approximately 45 minutes. Laser energy (1064 nm Nd:YAG) will be delivered via an optical fibre (300 μm core/320 μm clad) secured in a hand piece. Laser energy will be delivered by maintaining the tip of the optical fibre 3 mm from the treatment area to achieve around 1-1.5 mm diameter spot size (25.5 J/cm2 fluence per pulse; 10-pulse pulse-train to each spot in 0.5 seconds). Multiple treatment spots will be delivered to cover the entire area of involvement.
  Interventions: Device: Laser Treatment YAG laser
- Standard Treatment (control group) (Active Comparator): Control group volunteers will be asked to dedicate the same amount of time to the project with the same number of visits. However, they will receive conventional terbinafine therapy instead of laser treatments. Therefore, each of the 3 treatment visits would last only about 20 minutes.
  Interventions: Drug: Standard Treatment (control group) terbinafine hydrochloride tablets

INTERVENTIONS:
Device: Laser Treatment YAG laser — YAG Laser / FOX Laser
  Other Names: 1064 nm Nd:YAG laser; FOX laser
  Arms: Laser Treatment
Drug: Standard Treatment (control group) terbinafine hydrochloride tablets — Terbinafine hydrochloride tablets tablets
  Other Names: terbinafine hydrochloride tablets
  Arms: Standard Treatment (control group)

SUMMARY:
Fungal infections of the toe affect one in three people with diabetes. Current treatments for fungal toe infections include oral medications, but these drugs often interact with other common medications. We are studying a new treatment for fungal toe infections involving the use of a laser device. We will compare to the standard treatment which is a type of antifungal medication. This laser has been tested in small numbers of patients with minimal side effects. There will be 60 participants selected for our study, of which 30 will receive standard treatment and the rest will receive laser treatment.

DETAILED DESCRIPTION:
Onychomycosis is a fungal infection of the nail unit which affects one third of people with diabetes.1,2 Risk factors for onychomycosis in diabetes include age, male sex, poor glycemic control, longer duration of diabetes, use of immunosuppressive agents, and poor peripheral circulation.2-5 Etiology of onychomycosis varies across populations, but the most common causes in diabetic patients are yeasts and dermatophytes. In particular, Candida spp. (31-48.1%) are the most common yeasts, while Rhodotorula spp. (21.7%) have been reported as well.4,6-8 Trichophyton rubrum (31.7-46%) is the most common dermatophyte observed, while nondermatophytic molds are less common.

Individuals with diabetes complicated by peripheral neuropathy are at risk of developing particularly severe complications of onychomycosis. Infected nails can become brittle and sharp, injuring and compromising the adjacent skin. This breakdown allows a portal of entry for bacteria, causing cellulitis and paronychia.9 Because the nail bed is in close proximity to the underlying nail, paronychia can develop into osteomyelitis if adequate foot care is neglected.

Given the significant morbidity of onychomycosis including the potential for limb amputation, prompt and effective treatment is imperative. Currently available treatments include topical and systemic options, and each of these has significant limitations.

Topical antifungal therapies have been tested in patients with mild onychomycosis. Cure rates of 29-85% have been observed with ciclopirox 8% nail lacquer in non-diabetic populations with mild disease;10 in diabetic populations using open label methodology cure rates of approximately 54% are reported.11,12 Novel topical forms of terbinafine with various penetration-enhancing compounds are also under development.13-15 Early studies report effective nail penetration of these formulations, but there is a lack of data on clinical efficacy of topical terbinafine. One preliminary study reported 90% mycological cure after 12 weeks of treatment with a terbinafine spray, but less than half had a sustained cure at 36 weeks post-treatment.16 Although effective for mild to moderate superficial onychomycosis, because of poor nail penetration topical agents are generally not recommended where fungus appears to infect more than 50% of the nail surface.7 One recent review has suggested that monotherapy with topical agents should be avoided altogether.17 Systemic antifungal agents are often used to treat more severe onychomycosis. Two of the most common systemic agents are itraconazole and terbinafine. Itraconazole is a newer agent with the added advantage of covering Candida species in addition to dermatophytes. Both agents are associated with cure rates of approximately 50% when given for a full three month course.18 These agents have significant limitations given the potential for drug-drug interactions via inhibition of cytochrome P450 enzyme subtypes.19 Itraconazole and terbinafine are associated with increased risk of bleeding with warfarin, itraconazole with increased risk of rhabdomyolysis with statins and of hypoglycemia with oral agents for diabetes and terbinafine with metoprolol, propafenone, and tricyclic antidepressants.19 Due to the significant limitations of topical and systemic treatments for onychomycosis, there is a critical need for alternative and replacement therapies. While surgical techniques such as avulsion and nail plate removal can be employed for severe and resistant infections, these treatments are quite invasive and painful.7,20 Other device-based therapies for onychomycosis include UV light therapy21-23 and photodynamic therapy.24-27 While these modalities show evidence of in vitro efficacy, there have been no robust studies conducted yet that demonstrate any clinical effectiveness.

A promising device-based therapy is laser treatment. The neodymium-doped yttrium aluminum garnet (Nd:YAG) device emits a laser in a continuous or pulsed fashion, and the 1064 nm wavelength is thought to be optimal due to its ability to penetrate deeply into the nail bed to eradicate fungal growth.28 Although this device is approved by the US Food and Drug Administration for use in patients with onychomycosis for a "temporary increase in clear nail,"28 there is a lack of research demonstrating effectiveness beyond several pilot studies. One study demonstrated mycologic cure in 7 out of 8 patients with no major side effects aside from temporary nail discoloration and occasional pin prick sensation.29 The parameters for the laser included a 0.65 ms pulse duration, 2 mm spot size and 223 J/cm2 energy fluence, and treatment consisted of 2 to 3 sessions spaced at least 3 weeks apart. A Chinese study of 33 patients demonstrated a 51% to 53% cure rate in patients treated for eight and four sessions respectively, spaced at 1 week intervals using a 30 ms pulse duration and 3 mm spot size laser at 240-324 J/cm2.30 Results from Japan showed a similar cure rate of 51% in 19 patients treated with 1 to 3 treatments 4 to 8 weeks apart.31 To our knowledge, no randomized control trials exist to validate these preliminary findings.

Study Objectives The objective of this study is to determine the relative safety and clinical efficacy of laser treatment using the FOX Nd:YAG 1064 nm device compared to conventional therapy (topical terbinafine) in diabetics with onychomycosis of the hallux (great toe). Specifically, the study will test the hypothesis that participants randomized to the FOX Nd:YAG laser are more likely to be cured 6 months after initiating therapy compared to those randomized to conventional therapy. A secondary objective will be to determine the improvement in quality of life with laser treatment versus conventional therapy.

Subjects Eighty participants will be randomized equally to either the laser treatment group or the standard care group.

Study overview

This is a prospective, randomized, intention-to-treat, non-blinded comparative group clinical trial of 80 participants receiving laser or conventional, topical medication, therapy on a single infected hallux. All participants will have a baseline and 6 month follow-up visit where photographs of the hallux and repeat KOH and culture will be performed.

Participants randomized to laser group will undergo laser treatment at baseline and be asked to return for 2 subsequent visits six weeks apart (at weeks 6 and 12) to undergo further laser treatment of the hallux. Each visit will last approximately 45 minutes.

At the 6-month visit, participants randomized to the control group will be offered the first of three laser treatments (the second and third to occur at weeks 30 and 36). Participants in the laser group with persistent infections after 6 months will be offered standard therapy. No further data will be collected after the final 6-month visit.

The treatments will be performed at BCDiabetes (400 - 210 West Broadway, Vancouver, V5Y 3W2, Canada) owned and operated by Dr. Elliott .

Primary outcome measures One primary outcome will be the proportion of participants with microbiological cure (by KOH and culture) by 6 months post-randomization (i.e.: initiation of treatment).

Other primary outcomes include safety outcomes. Specifically, safety outcomes of interest will include the side effects listed below:

Usual side effect:

Feeling of warmth, heat, or tingling at the laser target site (only during treatment)

Rare side effects:

Discoloration/burn marks on surface of the nail Slight or mild pain (only during treatment) Redness of the treated skin around the nail (lasting 24-72 hours)

Rare laser effect:

Sometimes the laser creates 'sparks' on the surface of the nail - this does not cause any problems

Extremely rare laser effects Blistering of the treated skin around the nail Scarring of the treated skin around the nail

Secondary outcome measures Secondary outcomes will include the proportion of participants experiencing clinical cure by visual assessment (planimetry and photograph) will be evaluated.

The other secondary outcome will be improvement in quality of life as measured by the validated "NailQoL" questionnaire which assesses symptom, emotion, and functional domains.

Recruitment Patients ostensibly meeting the study inclusion and exclusion criteria seen in an outpatient setting by the authors and their associates and staff will be apprised of the availability of a research treatment for fungal toenail infection. The study will be briefly described - patients who express an interest will be provided additional information and a study consent form and be encouraged to ask questions about the study. They may choose to provide consent at the time or to leave with the consent form and return at a later time to ask further questions.

The anticipated accrual will be 80 patients in total. Screening Patients will participate in a screening visit as part of routine care. Informed consent will be obtained before any screening procedures. During this visit, toenail clippings will be sent for KOH stain and fungal culture. The results of these tests will be available in approximately 4 weeks. The results will be reviewed 6 weeks after the clippings are collected, and if the results are negative the patient will be excluded from study.

Patients positive for both KOH and fungal culture will be eligible for further screening with both ankle-brachial index evaluation and biothesiometry, and this screening would occur during the same visit.31-33 Patients with an ankle-brachial index less than 0.6 or biothesiometry score of less than 20 volts in either lower extremety will be excluded from participation as described in the exclusion criteria.

Samples will be collected only from the infected hallux, and if the hallux from both feet appear to be infected, samples from both feet will be taken and sent for analysis. If both right and left hallux samples are positive, one hallux will be chosen at random to be treated as part of the study.

Intervention Group Treatment Procedures

Laser energy (1064 nm Nd:YAG) will be delivered via an optical fibre (300 μm core/320 μm clad) secured in a hand piece. Laser energy will be delivered by maintaining the tip of the optical fibre 3 mm from the treatment area to achieve around 1-1.5 mm diameter spot size (25.5 J/cm2 fluence per pulse; 10-pulse pulse-train to each spot in 0.5 seconds). Multiple treatment spots will be delivered to cover the entire area of involvement. Treatments cause no discomfort and are administered as an outpatient service with no anesthesia. If the subject experiences significant discomfort, the procedure may be interrupted for up to 5 minutes to allow the discomfort to subside.

The FOX laser will be used in accordance with manufacturer recommendations, with output power, spot size, and proprietary pulse train incorporated into the treatment regimen. Treatment will take place by traversing the infected hallux in a side to side fashion, with care being taken to cover the entire surface of each nail, by slightly overlapping the previous path. In areas where the nail appears to be infected, a second series of passes perpendicular to the first set will be performed, again slightly overlapping the previous path, as described above. Even if other toes in addition to the hallux appear to be infected, only one hallux per participant will be treated and analyzed for the purposes of the study. The treatment will be performed as an outpatient procedure at St. Paul's Hospital or Mount St. Joseph's Hospital.

Participants who fail to return for a scheduled treatment will be asked to return for another treatment as soon as possible. The schedule for subsequent treatments will be readjusted based on the completion date of the missed visit.

Control Group Treatment Procedures

Participants in the control group will be treated conventionally with terbinafine HCl external ointment.

Planimetry Procedures

Photographic documentation and assessment of the treated toenails will be done at the interval visits as listed in the subject follow-up table below. The extent of mycological involvement will be determined by measuring the mm of clear nail from the cuticle line to the demarcation of clinically involved nail. This data will be recorded in the case report form. Nails are scored (grooved) at the initial visit to indicate the most proximal level of involvement. The distance from the proximal cuticle to the scored mark will be measured at each visit on any involved hallux nail.

The photograph will be analyzed using ImageJ software version 1.4.1 ( HYPERLINK "http://rsb.info.nih.gov/ij/docs/intro.html"http://rsb.info.nih.gov/ij/docs/intro.html), a public domain Java image processing program inspired by NIH Image written by Wayne Rasband ( HYPERLINK "mailto:wayne@codon.nih.gov"wayne@codon.nih.gov), Research Services Branch, National Institute of Mental Health, Bethesda, Maryland, USA. The software will be used by an expert PathoLase photo-evaluator to measure the linear distance of non-involved toenail (e.g., clear of infection) immediately before treatment (baseline) and 6 months.

Withdrawal and End of Participation

A participant is free to withdraw from the study at any time, for any reason without prejudice to their future medical care by the physician or at the institution. The Investigator also has the right to withdraw participants from the study in the event of intercurrent illness, adverse events, administrative, or other reasons unrelated to the study if such a decision is in the subject's best medical interest.

When a participant withdraws from the study, all assessments required at the 6-month study visit will be obtained, where possible. All details available will be reported and recorded for any subject who withdraws from the study. Participants, who wish to withdraw from treatment, will be encouraged to return for their 6-month study visit to complete the required examination.

If a participant is lost to follow-up, at least 3 documented attempts must be made to contact the subject, one of which must include sending a certified letter to the participant's last known address, which includes a request to return to the study site for final study evaluations.

Participants who fail to return for their 6-month visit will be considered failures (i.e. no microbiological cure) unless a nail clippings were obtained from a prior visit and confirmed as microbiological cure.

Information on whether microbiological cure was achieved during the study will be shared with subjects as well as their health care providers.

At the completion of study procedures, laser treatment will be offered to control group participants as well as to intervention group participants who wish to have additional toes treated.

Risks and Discomforts The following is a list of risks and possible discomforts associated with the FOX Nd:YAG 1064 nm laser. Precise estimates of the percentage occurrence of these side effects are not available given the limited number of pilot studies available.

Usual side effect:

Feeling of warmth, heat, or tingling at the laser target site (only during treatment

Rare side effects:

Discoloration/burn marks on surface of the nail Slight or mild pain (only during treatment) Redness of the treated skin around the nail (lasting 24-72 hours)

Rare laser effect:

Sometimes the laser creates 'sparks' on the surface of the nail - this does not cause any problems

Extremely rare laser effects (did not occur during clinical studies):

Blistering of the treated skin around the nail Scarring of the treated skin around the nail

Significant side effects were not reported in several small pilot studies of the Nd:YAG 1064 nm laser. We will minimize the risk of side effects by using the laser strictly according to the manufacturer-recommended protocol described in the intervention section above. We would consider stopping the study early if severe side effects such as blistering and scarring are unexpectedly observed in a significant proportion of study participants.

Side effects for the control group receiving topical terbinafine are to be expected as part of the current standard of care. The known side effects of this conventional treatment are detailed as below:

Dermatologic side effects (1-10%): Burning, contact dermatitis, dryness, exfoliation, irritation, pruritus, rash Local side effects (1-10%): Irritation, stinging Statistical Analysis

Analysis Supporting the Primary Objective

The primary outcome measure is the proportion of participants with microbiological cure (by KOH and culture) by 6 months post-baseline treatment. The null and research hypotheses supporting the primary objective of investigating the impact of whether laser treatment, using the FOX Nd:YAG 1064 nm device, is more effective in the treatment onychomycosis in comparison to conventional therapy (topical terbinafine) is then:

H0: pc ≥ ptr vs. H1: pc < ptr where pc and ptr are the proportion of subjects with microbiological cure (by KOH and culture) by 6 months post-baseline treatment, within the control group, and the laser group respectively. Here, rejecting the null hypothesis implies that the proportion of participants achieving microbiological cure is higher in the laser group. A 1-sided, 0.05 alpha-level Fisher's exact test for proportions will be used.34

The rate of each safety outcome (feeling of warmth/heat/tingling, discolouration or burn marks, pain, redness, sparks, blistering, scarring), and accompanying 95% exact binomial confidence interval, will be calculated.

Sample Size Considerations

Based on previous studies, terbinafine may be associated with cure rates of approximately 50% (when given for a full three month course).18 The success rate of the FOX laser group has not been thoroughly investigated. Table 2 provides the power to detect various true differences between the control and laser groups where the control group is assumed to have a success rate between 40% and 60%. A sample size of 80 subjects in a 1:1 randomization to the control and laser arm will provide a power of 80% to reject the null hypothesis if the laser arm true cure rate in the control arm is 79% and the control arm is achieves a cure rate of 50%. If the success rate in the control group is as high as 60%, a difference of 26% between the groups will be detectable with 80%. If the true difference is 34% or greater, it will be detected with at least 90% power. For a total sample size of 100, a true difference of at least 31% will be detectable with at least 90% power, a reduction of only 3%. Similarly, for a total sample size of 60, the difference must be at least 39% to be detected with at least 90% power, an increase of 4%.

Human Subjects Protection This study will be conducted in accordance with the ethical principles originating from the Declaration of Helsinki and Good Clinical Practices (GCP) defined in ICH E6 and in compliance with provincial and national regulatory requirements.

Justification for exclusion of children

Justification for exclusion of other vulnerable subjects (Vulnerable subjects include who lack consent capacity, mentally ill, prisoners, cognitively impaired subjects, pregnant women, etc.

Justification of sensitive procedures Our study does not involve the use of placebo, medication withdrawal, provocative testing, or deception.

Safeguards for vulnerable populations:Females of childbearing potential must agree to practice sexual abstinence or use a medically acceptable method of contraception for the duration of the study and for at least 1 month after the last day of test article administration Anticipated Benefit Study participants randomized to the medication group will receive the current best available treatment for onychomycosis. Participants who fail to be cured by this treatment will have the option to undergo treatment with the laser following the 6 month study visit. It is possible that participants randomized to the laser treatment will be more likely to be cured than the standard treatment.

Consent documents and process All subjects for this study will be provided with a consent form describing this study and providing sufficient information for subjects to make an informed decision about their participation in this study. This consent form will be submitted with the protocol for review and approval by the REB for the study. The formal consent of a subject, using the REB approved consent form, must be obtained before that subject undergoes any study procedure. The consent form must be signed by the subject or by a legally acceptable surrogate, and the Investigator and/or designated research professional obtaining the consent. A copy of the signed and dated informed consent form must be given to the subject and the consent process must be documented.

Quality Assurance Before enrolling any subjects in this study, the Investigator and other staff will review the protocol, the source documents and instructions for their completion, the procedure for obtaining informed consent, and the procedure for reporting AEs and SAEs.

Collected data will be reviewed for completeness on a monthly basis and include a review of missing data elements, missing or out-of-window visits, and any other anomalies.

Adverse event and unanticipated problem reporting

Adverse Events

An adverse event (AE) can be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of an investigational product. The event does not need to be causally related to the test article or clinical study. An AE includes, but is not limited to, the following:

Any clinically significant worsening of a pre-existing condition. An AE occurring from overdose of a test article, whether accidental or intentional. Overdose is a dose greater than the dose (i.e. laser intensity) specified for each test article in section 4.2.

An AE occurring from abuse (e.g., use for nonclinical reasons) of a test article.

An AE that has been associated with the discontinuation of the use of a test article.

The severity of all adverse events is graded as follows:

Mild

Signs or symptoms, usually transient, requiring no special treatment and generally not interfering with usual activities

Moderate

Signs or symptoms, which may be ameliorated by simple therapeutic measures, may interfere with usual activity.

Severe

Signs or symptoms that are intense or debilitating and that interfere with usual activities. Recovery is usually aided by therapeutic measures and the discontinuation of the study device may be required.

The relationship of each adverse event to the study was defined as follows:

Probable

An adverse event has a strong temporal relationship to study device, and another etiology is unlikely or significantly less likely.

Possibly

An adverse event has a strong temporal relationship to the study device, and an alternative etiology is equally or less likely compared to the potential relationship to study device.

Not related

An adverse event has no temporal relationship to study device or has a much more likely alternative etiology.

Serious Adverse Events

A serious adverse event (SAE) is an AE that:

Results in death; Is life-threatening, i.e., an event that places the subject, in the view of the Investigator, at immediate risk of death from the event as it occurred (does not include an event that, had it occurred in a more severe form, might have caused death); Requires inpatient hospitalization or prolongation of an existing hospitalization; Results in persistent or significant disability or incapacity; Results in cancer; Results in a congenital anomaly or birth defect; Other medically important events that in the opinion of the Investigator may jeopardize the subject or may require intervention to prevent one of the other outcomes listed in the definition above; Any serious problem associated with the device that relates to the rights, safety or welfare of study subjects.

Reportable Incidents

According to the Canadian Medical Devices Regulations (Sections 59 and 81), a reportable incident is any incident that:

Is related to a failure of the device or a deterioration in its effectiveness, or any inadequacy in its labeling or in its directions for use; and Has led to the death or a serious deterioration in the state of health of a participant, user or other person, or could do so were it to recur.

Efficacy Endpoints and Disease Progression Event

In general, an event of treatment failure or lack of treatment efficacy is not considered an SAE. If, however, it results in a situation that qualifies as an SAE as defined above, it should be reported. Treatment failure/lack of efficacy will be captured on the clinical evaluation source documents and, if it results in discontinuation of test article or withdrawal from the study, should be captured on those source documents as well.

Recording of Adverse Events

At each contact with the subject, the Investigator will seek information on adverse events by specific questioning and, as appropriate, by examination of the subject. Information on all adverse events should be recorded immediately. All clearly related signs, symptoms, and abnormal diagnostic procedure results should be recorded, though should be grouped under one diagnosis.

All adverse events occurring during the study period must be recorded. The clinical course of each event should be followed until resolution, stabilization, or until it has been determined that the study treatment or participation is not the cause.

Confidentiality

Information about study subjects will be kept confidential and managed according to the requirements of the Federal and Provincial Data Protection regulations, including the Personal Information Protection and Electronic Documents Act (PIPEDA 2000). Those regulations require signed subject authorization, informing the subject of the following:

What protected health information (PHI) will be collected from subjects in this study; Who will have access to that information and why; Who will use or disclose that information; The rights of a research subject to revoke their authorization for use of their PHI.

In the event that a subject revokes authorization to collect or use PHI, the Investigator, by regulation, retains the ability to use all information collected prior to the revocation of subject authorization. For subjects that have revoked authorization to collect or use PHI, attempts should be made to obtain permission to collect at least vital status (i.e. that the subject is alive) at the end of their scheduled study period.

Data Access

Data will be stored in electronic medical records within the clinical practice. Data will be accessed only by study investigators or the study statisticians. Individual level data will be identified only with study registration numbers.

Records Retention

The Investigator shall retain and preserve electronically all data generated in the course of the study, specifically including but not limited to those defined by GCP as essential for 25 years from the date of the completion of the study.

Conflict of Interest Study investigators have no financial interests relating to the laser or medication arms of these studies.

ELIGIBILITY:
Inclusion Criteria:

* Provides full informed consent to participate in the study;
* At least 19 years of age;
* Established diagnosis of diabetes mellitus at the time of screening for the study according to Canadian Diabetes Association (CDA) criteria;
* Clinically assessed to have subungual onychomycosis (fungal infection of the nail) of the hallux, confirmed by KOH and culture performed at the screening visit.

Exclusion Criteria:

* Presence of necrotizing fasciitis, cellulitis, wet gangrene, gas gangrene, erythema gangrenosum, or psoriasis;
* Presence of peripheral arterial disease defined as an ankle-brachial index less than 0.6 on either lower extremity;
* Presence of peripheral neuropathy defined as a biothesiometry score of less than 20 volts on either lower extremity;
* Treatment with oral terbinafine (Lamisil), itraconazole (Sporanox), or griseofulvin within 12 months of the proposed study start date;
* Treatment with any topical antifungal medications including ciclopirox, itraconazole, or other over-the-counter remedies for toenail infection within 1 month of randomization;
* Female of childbearing potential who does not agree to practice sexual abstinence or use a medically acceptable method of contraception for the duration of the study and for at least 1 month (30 days) after the last day of test article administration; (A woman of childbearing potential is one who is biologically capable of becoming pregnant; this includes women who are using contraceptives or those women whose sexual partners are either considered sterile or using contraceptives.)
* Has a physical disability or psychiatric diagnosis which would limit the ability to adhere to the study regimen, as judged by the Investigator;
* Is a prisoner, or is in pre-trial;
* Is known to be without a fixed address;
* Has documented evidence of a history (e.g. liver testing) of substance abuse within the 12 months prior to screening for study entry;
* Is a Workers Compensation Board (WCB) patient;
* Is unable to easily communicate in oral and written English.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Microbiological Cure | 6 months
  One primary outcome will be the proportion of participants with microbiological cure (by KOH and culture) by 6 months post-randomization (i.e.: initiation of treatment).
Side effects from laser treatment | 6 months
  Other primary outcomes include safety outcomes. Specifically, safety outcomes of interest will include the side effects listed below:
  * Usual side effect:
    o Feeling of warmth, heat, or tingling at the laser target site (only during treatment)
  * Rare side effects:
    * Discoloration/burn marks on surface of the nail
    * Slight or mild pain (only during treatment)
    * Redness of the treated skin around the nail (lasting 24-72 hours)
  * Rare laser effect:
    o Sometimes the laser creates 'sparks' on the surface of the nail - this does not cause any problems
  * Extremely rare laser effects:
    * Blistering of the treated skin around the nail
    * Scarring of the treated skin around the nail

SECONDARY OUTCOMES:
Clinical cure by visual assessment | 6 months
  Secondary outcomes will include the proportion of participants experiencing clinical cure by visual assessment (planimetry and photograph) will be evaluated.
Quality of Life | 6 months
  The other secondary outcome will be improvement in quality of life as measured by the validated "NailQoL" questionnaire which assesses symptom, emotion, and functional domains.38

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Elliott, MBBS, Principal Investigator — University of British Columbia
Locations (1):
- Diamond Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
There is no initial plan to share IPD at the moment

REFERENCES:
- [Background] Ledon JA, Savas J, Franca K, Chacon A, Nouri K. Laser and light therapy for onychomycosis: a systematic review. Lasers Med Sci. 2014 Mar;29(2):823-9. doi: 10.1007/s10103-012-1232-y. Epub 2012 Nov 20. PMID 23179307
- [Background] Hochman LG. Laser treatment of onychomycosis using a novel 0.65-millisecond pulsed Nd:YAG 1064-nm laser. J Cosmet Laser Ther. 2011 Feb;13(1):2-5. doi: 10.3109/14764172.2011.552616. Epub 2011 Jan 21. PMID 21250792
- [Background] Zhang RN, Wang DK, Zhuo FL, Duan XH, Zhang XY, Zhao JY. Long-pulse Nd:YAG 1064-nm laser treatment for onychomycosis. Chin Med J (Engl). 2012 Sep;125(18):3288-91. PMID 22964325
- [Background] Kimura U, Takeuchi K, Kinoshita A, Takamori K, Hiruma M, Suga Y. Treating onychomycoses of the toenail: clinical efficacy of the sub-millisecond 1,064 nm Nd: YAG laser using a 5 mm spot diameter. J Drugs Dermatol. 2012 Apr;11(4):496-504. PMID 22453588